CLINICAL TRIAL: NCT04957472
Title: Multicenter Study of the Safety and Performance of Fabian-PRICO for Saturation Targeting Routine Use in the NICU
Status: Completed | Type: Observational
Sponsor: Vyaire Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 21-001-PRICO
Record Dates: First submitted 2021-06-30; First posted 2021-07-12 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Respiratory Insufficiency in Children

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

INTERVENTIONS:
Device: fabian HFO, fabian +nCPAP evolution and fabian Therapy evolution with PRICO function — 24 hours of automated control of FiO2
Other: Manual Control — 24 hours of manual control of FiO2

SUMMARY:
This study is planned as a part of the post market clinical follow-up (PMCF) on a CE marked product. The purpose of the study is to demonstrate, in a routine clinical environment across a number of centers, that the fabian-PRICO can adequately maintain oxygen saturation, with minimal staff intervention.

DETAILED DESCRIPTION:
This is a randomized cross-over study. Subjects will be assigned to two, nominally 24-hour interventions, one with standard manual titration of FiO2 and the other with automated adjustment (PRICO). The order of these two interventions will be random.

In addition to the ventilators data, basic demographics (i.e., gestational age, birth weight, age, weight at study) of the participating infants will be recorded in the eCRF.

This study has no additional follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Respiratory insufficiency of infants in the neonatal unit who require respiratory support and supplemental oxygen in one of 4 the therapeutic categories (Intubated HFO, Intubated CMV, Non-Invasive nasal mask, nasal cannula).
* <30 kg at study entry
* Informed Consent Form obtained as per EC requirement

Exclusion Criteria:

* Not expected to complete 48 hours of the current respiratory support therapeutic category
* Congenital anomalies
* Uncontrolled hemodynamics
* Severe airflow obstruction
* Intracranial hypertension
* Start of caffeine therapy within 12 hours
* Attending physician does not believe participation of the patient is in their best interest.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Members of the Investigational team will periodically review records to identify and maintain a pool of potential investigation candidates from the NICU. It is anticipated that this pool will be significantly larger than capacity of the team to enroll into the investigation.
  The parents of potential candidates will be approached for discussion and consent prior to the desired intervention.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Target Range Compliance: | 24 hours
  Percent-Time with SpO2 a) <80% and b) with >98% SpO2 with FiO2>21%

SECONDARY OUTCOMES:
Avoidance of SpO2 Extremes: | 24 hours
  Percent-Time with SpO2 a) <80% and b) with >98% SpO2 with FiO2>21%

CONTACTS AND LOCATIONS:
Overall Officials: Maria Wilińska, MD, PhD, Principal Investigator — Centre of Postgraduate Medical Education, SPSK im prof.W.Orłowskiego Warsaw; Anton HLC van Kaam, Prof. MD PhD, Principal Investigator — University Medical Center, Amsterdam, The Netherlands
Locations (5):
- Amsterdam UMC, Amsterdam, Netherlands
- Poland (4):
  - Szpital Położniczo - Ginekologiczny Ujastek, Krakow
  - Ginekologiczno-Położniczy Szpital Kliniczny Uniwersytetu Medycznego im. K. Marcinkowskiego, Poznan
  - SPSK 2 Pomeranian Medical University, Szczecin
  - Centre of Postgraduate Medical Education, SPSK im prof.W.Orłowskiego Warsaw, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wilinska M, Bachman T, Szczapa T, Wroblewska-Seniuk K, Chojnacka K, Loniewska B, Olszanska K, Rzepecka Weglarz B, Janusz K, Piwowarczyk P, Onland W, Hutten GJ, van Leuteren RW, van Kaam AH. Performance and safety of the PRICO closed-loop oxygen saturation targeting system in neonates: pragmatic multicentre cross-over study (TarOx Study). BMJ Paediatr Open. 2024 Jul 16;8(1):e002583. doi: 10.1136/bmjpo-2024-002583. PMID 39019542
- See also: Performance and safety of the PRICO closed-loop oxygen saturation targeting system in neonates: pragmatic multicentre cross-over study (TarOx Study) — https://pubmed.ncbi.nlm.nih.gov/39019542/